CLINICAL TRIAL: NCT06016569
Title: Prospective Validation Study of Early Cancer Biomarkers in Breath Condensate of Individuals With High-Risk of Lung Cancer Undergoing Low-Dose Computer Tomography Based Screening.
Brief Title: Study of Early Cancer Biomarkers in Breath Condensate in Population of Individuals With High-Risk of Lung Cancer Undergoing LDCT Screening.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: Cancer Research Foundation CR (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 60096
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Breath Condensate; Biomarker; Screening; Early Cancer Detection
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Vital Signs; Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDCT and collection of breath condensate and blood sample (Experimental): Each participant of the study will provide exhaled breath condensate sample and blood sample for further laboratory analyses. Each participant will have LDCT (low dose computer tomography) performed. A pulmonologist examines the patient for any concomitant diseases and performs spirometry. Vital signs will be measured.
  Interventions: Diagnostic Test: Exhaled breath condensate sampling; Diagnostic Test: Blood sampling; Procedure: LDCT; Diagnostic Test: Vital signs; Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Exhaled breath condensate sampling — Patient will breath for approx. 10 minutes to a breath condenser. The exhaled breath sample will be condensed and freezed.
Diagnostic Test: Blood sampling — A venous blood sample will be taken for further biomarker analysis.
Procedure: LDCT — LDCT scan will be performed.
  Other Names: Low Dose Computer Tomography
Diagnostic Test: Vital signs — Blood pressure, weight, height, pulse, oxygen saturation will be measured.
Diagnostic Test: Spirometry — Spirometry will be performed.

SUMMARY:
The trial will evaluate if the newly identified biomarkers of lung cancer in exhaled breath condensate are as a diagnostic tool comparable to the low-dose computer tomography (LDCT) implemented in lung cancer screening recently. Due to the possibility to collect breath condensate at any medical workplace and due to the relatively low financial cost of examination of the collected breath condensate could improve early diagnosis of lung cancer, differential diagnostics of lung nodules and thereby reduce both the unnecessary interventions and deaths from this type of cancer.

DETAILED DESCRIPTION:
The project aims to validate newly identified biomarkers of lung cancer in breath condensate for the diagnosis and triage of lung nodules (malignant versus benign), further set the mechanisms of the functioning of the lung cancer screening center, validate the quality indicators of LDCT screening for the Czech Republic and stratify the cohort of individuals so that optimized output of screening activities. Patients aged 55-74 years with a heavy smoking load (more than 20, preferably more than 30 pack/years) will be divided into risk groups according to biomarkers in exhaled air, clinical/anamnesis data and the degree of obstructive ventilation disorder according to spirometry and subsequently there will be effective stratification of the risk of lung carcinoma. The group with the highest risk of developing lung cancer will then be diagnosed with early lung cancer using ultra-low-dose computed tomography of the chest. This will lead to early diagnosis and subsequently to a reduction in the mortality rate of the monitored active group compared to the historical cohort. The primary outcome will be the validation of the multiplex protein signature in exhaled air, the effectiveness of the screening procedure to reduce lung cancer mortality and overall mortality in the group with FEV1 (forced expiratory volume at 1 second) pre-bronchodilation 60-75% with the entire group of examinees. The secondary outcome will then be the total time of diagnosis of a solitary pulmonary nodule in positively screened patients for whom only observation is not a sufficient procedure. Another secondary outcome will be the costs of screening procedures for individual groups and the percentage of success of the anti-smoking intervention for the enrolled individuals. The number of newly captured interstitial lung processes will also be evaluated. Patients will be evaluated for 5 years at annual visits or earlier based on their LDCT result.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in a clinical trial.
2. A clients within an age of 55-74 years.
3. Current smoker or ex-smoker who has smoked at least 20 pack-years, provided that:

   1. priority will be given to clients who have smoked at least 30 pack-years.
   2. preference will be given to a former smoker who has not smoked for less than 15 years.

Exclusion Criteria:

1. Previous diagnosis of lung cancer.
2. Progressing malignant tumor on symptomatic treatment.
3. Advanced dementia
4. Chronic obstructive pulmonary disease or other inflammatory disease in the phase of acute exacerbation.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Validation of the multiplex protein signature in exhaled air | 5 years
  Validation of the multiplex protein signature in exhaled breath condensate based on the comparison with the LDCT.
Validation of the multiplex protein signature in exhaled breath for differential diagnostics of lung nodules | 5 years
  Validation of the multiplex protein signature in exhaled breath for differential diagnostics of lung nodules
Assessment of the effectiveness of the screening program | 5 years
  Assesment of the effectiveness of the screening procedure to reduce lung cancer mortality and overall mortality in the group with FEV1 (forced expiratory volume at 1 second) pre-bronchodilation 60-75% compared with the entire group of examinees.

SECONDARY OUTCOMES:
Total time of diagnosis of the nodule | 5 years
  The total time of diagnosis of a solitary pulmonary nodule in positively screened patients for whom only observation is not a sufficient procedure.
Comparison of costs of screening procedures | 5 years
  Comparison of the costs of the screening procedures for exhaled breath condensate sample and LDCT procedure. This will be asssessed based on the individula patient data: total screening costs per patient from Healthcare registry in Czech Republic.
Assessment of success of the anti-smoking intervention | 5 years
  Percentage success of the anti-smoking intervention in the examined probands.

OTHER OUTCOMES:
Number of newly captured interstitial lung processes | 5 years
  The number of newly captured interstitial lung processes will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD, PhD., Study Director — IMTM, Palacky University in Olomouc, Faculty of Medicine and Dentistry
Locations (3):
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital, Olomouc
  - General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No